CLINICAL TRIAL: NCT06889012
Title: An Open-label, Randomized, Fasting, Single-dose, 2-sequence, 4-period, Crossover Phase 1 Study to Evaluate the Pharmacokinetics and the Safety After Administration of "BR1018" and Coadministration of "BR1018A" and "BR1018B" in Healthy Volunteers
Brief Title: A Study to Evaluate the Pharmacokinetics and the Safety After Administration of BR1018 and Coadministration of BR1018A and BR1018B in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-FAEAC-CT-103
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Essential Hypertension; Primary Hypercholesterolemia
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BR1018 (Experimental)
  Interventions: Drug: BR1018
- BR1018A+BR1018B (Active Comparator)
  Interventions: Drug: BR1018A; Drug: BR1018B

INTERVENTIONS:
Drug: BR1018 — One tablet administered alone
  Arms: BR1018
Drug: BR1018A — One tablet administered alone
  Arms: BR1018A+BR1018B
Drug: BR1018B — One tablet administered alone
  Arms: BR1018A+BR1018B

SUMMARY:
The purpose of this clinical study is to evaluate the pharmacokinetics and the safety after administration of BR1018 and coadministration of BR1018A and BR1018B in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Those who have body mass index (BMI) of more than 18.0kg/m2 and less than 30.0kg/m2 at screening visit.

  * For men, Those who weigh 50 kg or more
  * For women, Those who weigh 45 kg or more
* Those who sign written consent spontaneously after listening to and understanding sufficient explanation of the purpose and contents of this clinical trial, characteristics of the Investigational products, expected adverse events, etc.
* Those who agree to rule out the possibility of their and their spouses' or sexual partners' pregnancy by using methods of contraception accepted in clinical trial*(Except for hormone drugs) from the date of consent to 14 days after the last administration and disagree to provide their sperm or ovum.

  * Methods of contraception accepted in clinical trial: Combined use of intrauterine device, vasectomy, tubal ligation, and barrier methods (male condom, female condom, cervical cap, contraceptive diaphragm, sponge, etc.) or combined use of two or more barrier methods if spermicide is used.

Exclusion Criteria:

* Those who have taken drugs that induce and inhibit metabolizing enzymes such as barbiturate within 30 days before the first administration date or have taken drugs concerned about affecting this clinical trial within 10 days before the first administration date. (However, participation is possible considering pharmacokinetics and pharmacodynamics such as Interaction of investigational products, half-life of concomitant drugs, etc.)
* Those who have a medical history of gastrointestinal resection or gastrointestinal diseases that may affect the absorption of drugs. (Except for simple appendectomy, hernia surgery)
* Those who have participated in other clinical trials(including bioequivalence tests) and administered their investigational products within 6 months before the first administration date. (However, the termination for participation in other clinical trials are based on the last administration date of their investigational products)
* Those who can't discontinue a diet (ex. raw grapefruit, grapefruit juice or food containing grapefruit, etc.) that may affect the absorption, distribution, metabolism, and excretion of the drug within 48 hours before the first administration date
* In the case of a female subject, those suspected pregnancy or pregnant woman or lactating woman.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-05-07 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
AUCt | 0-72 hours after administration
  Area under the plasma drug concentration-time curve from 0 to time t
Cmax | 0-72 hours after administration
  Maximum concentration of drug in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, H PLUS Yangji Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No